CLINICAL TRIAL: NCT02933658
Title: Study of Multiple Oral Dosing to Evaluate the Safety and the Pharmacokinetic Drug-drug Interaction of Telmisartan/Amlodipine and Rosuvastatin in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DW-1501-P101
Record Dates: First submitted 2016-10-12; First posted 2016-10-14 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Hypertension and Dyslipidemia
MeSH Terms: conditions — Hypertension; Dyslipidemias | interventions — Telmisartan; Amlodipine; Rosuvastatin Calcium

ARMS (2):
- Reference1 (Experimental): single(Reference1) -> combination(Reference1+Reference2)
  Interventions: Drug: Telmisartan; Drug: Amlodipine; Drug: Rosuvastatin
- Reference2 (Experimental): single(Reference2) -> combination(Reference1+Reference2)
  Interventions: Drug: Telmisartan; Drug: Amlodipine; Drug: Rosuvastatin

INTERVENTIONS:
Drug: Telmisartan
Drug: Amlodipine
Drug: Rosuvastatin

SUMMARY:
A non-randomized, two-arm, single-sequence, crossover, open label, multiple oral dosing clinical trial to evaluate the safety and the pharmacokinetic drug-drug interaction of Telmisartan/Amlodipine and Rosuvastatin in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male who are ≥19, <50 years old
* Man who weights over 55kg and whose BMI is 18~30(kg/m2)
* Man who doesn't have any chronic disease or history of disease

Exclusion Criteria:

* man who has or had any clinically relevant disease of liver, kidney, nervous/respiratory/musculoskeletal/cardiovascular/hemato-oncology system or neuropsychiatry

Ages: 19 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2015-11; Primary Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
AUC of Reference 1 | 0, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24hour
Cmax of Reference 1 | 0, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24hour
AUC of Reference 2 | 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24hour
Cmax of Reference 2 | 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24hour